CLINICAL TRIAL: NCT01885793
Title: Cuff Pressure in Patients: Manometer vs Invasive Pressure Monitoring Setup
Status: Completed | Type: Observational
Sponsor: Senthil G. Krishna (Other)
Responsible Party: Sponsor-Investigator, Senthil G. Krishna, Assistant Clinical Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00107
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Anesthesia Intubation Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cuffed endotracheal tube: Surgical patients who require endotracheal intubation with a cuffed endotracheal tube (ETT).
  Interventions: Device: Cuffed endotracheal tube

INTERVENTIONS:
Device: Cuffed endotracheal tube — Intubation with a cuffed endotracheal tube (ETT).

SUMMARY:
This is a prospective study looking at ways to measure the cuff pressure of cuffed endotracheal tubes (ETTs). We will be comparing a hand-held manometer (MM) to the transducer of an invasive pressure monitoring setup (IPMS), which is commonly used for arterial or central venous pressure monitoring. The investigators previously did this study in vivo with ETTs in polyvinyl chloride (PVC) "tracheas" and we found that there is good correlation between the pressure readings using the MM and the IPMS. The purpose of the current study is to validate the in vitro findings in clinical situations.

ELIGIBILITY:
Inclusion Criteria:

* Intubation of trachea with a cuffed endotracheal tube.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgical patients that require endotracheal intubation.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Intracuff pressure | Immediately after intubation
  Intracuff pressure is measured via handheld manometer and by using the transducer of an invasive pressure monitoring device.

CONTACTS AND LOCATIONS:
Overall Officials: Senthil Gopalakrishnan, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States